CLINICAL TRIAL: NCT05438056
Title: The Effect of the Mobile Application Developed for Home Care of the Premature Baby on the Mother's Baby Care Skills, Self-efficacy and Mother-infant Bonding
Brief Title: The Effect of the Mobile Application Developed for Home Care of Preterm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Gülçin KORKMAZ YENİCE, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraU06GKY
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Mother; Premature; Education; Home Care; Mobile Application
Keywords: Mothers, premature, mobile application, education, home care
MeSH Terms: conditions — Premature Birth | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: randomized controlled interventional research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- providing training to mothers of premature babies with a mobile application (Experimental): providing training with mobile application to mothers discharged home with their premature babies +standard education prior to discharge
  Interventions: Other: education with mobile application
- standard education prior to discharge control group; standard education prior to discharge (No Intervention): standard education prior to discharge

INTERVENTIONS:
Other: education with mobile application — providing training to mothers of premature babies with a mobile application
  Arms: providing training to mothers of premature babies with a mobile application

SUMMARY:
mobile application will be developed to support the post-discharge home care of mothers of premature babies. With the developed mobile application, the effect of the education given to the mothers on the knowledge and skills of infant care, mother-infant attachment, and the mother's self-efficacy will be evaluated.

DETAILED DESCRIPTION:
This research aims to examine the effect of the mobile application developed for the home care of the babies of the mothers of premature babies on their baby care knowledge and skills, mother-infant attachment and mother self-efficacy. A mobile application will be developed to support mothers who care for their premature babies at home after discharge. The application will be installed on the phones of mothers whose babies are discharged from the neonatal intensive care unit. After the babies are discharged, mothers will be trained at home with a mobile application. Maternal self-efficacy and mother-infant supplementation will be measured when infants admitted the NICU and one month after discharge the NICU.

ELIGIBILITY:
Inclusion Criteria:

For mothers;

* Being over the age of 18,
* Having a premature baby
* At least primary school graduate,
* Smart mobile app can be installed have a phone,
* Being able to understand and speak Turkish,
* Residing in Ankara

For babies;

* 32-37 weeks of gestation of the baby (middle and borderline premature)
* Baby in neonatal intensive care unit to stay
* Not having undergone a surgical operation,
* Absence of physical anomalies

Exclusion Criteria:

For Mothers;

* Diagnosed with postpartum depression
* unwillingness to participate in the study

For babies;

- Very small preterm (born below 28 weeks of gestation) and small preterm (between 28 and 31 weeks of gestation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-16 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
parent self-efficacy scale | up to 10 months
  scale that measures mother's self-efficacy for baby care.The unabridged name of the scale is parent self-efficacy scale. The lowest score obtained from the scale is 18, the highest score is 90. low score indicates high self-efficacy
parent self-efficacy scale | up to 14 months
  scale that measures mother's self-efficacy for baby care.The unabridged name of the scale is parent self-efficacy scale. The lowest score obtained from the scale is 18, the highest score is 90. low score indicates high self-efficacy.

SECONDARY OUTCOMES:
maternal attachment scale | up to 10 months
  scale that measuring mother-infant attachment. The unabridged name of the scale is maternal attachment scale. The lowest score obtained from the scale is 26, the highest score is 104. A high score indicates high maternal attachment.
maternal attachment scale | up to 14 months
  scale that measuring mother-infant attachment. The unabridged name of the scale is maternal attachment scale. The lowest score obtained from the scale is 26, the highest score is 104. A high score indicates high maternal attachment.

OTHER OUTCOMES:
baby care knowledge and skills form | up to 14 months
  Form that measuring baby care knowledge and skills. The unabridged name of the form is baby care knowledge and skills form. Since the form created by the researcher has not been finalized, the lowest and highest scores to be obtained from the form are not certain. A high score indicates a high level of knowledge and skill of the mother.

IPD SHARING:
Plan to Share IPD: No
When the study is completed and published, the score obtained from the parent self-efficacy scale and maternal attachment scale will be shared.